CLINICAL TRIAL: NCT06442969
Title: Implementing an Intervention to Reduce Heat Stress and Chemical Exposures
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: San Diego State University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HS-2024-0081
Record Dates: First submitted 2024-05-13; First posted 2024-06-05 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Dehydration; Heat Stress
Keywords: Farm worker; Heat exposure; Chemical exposure; Agricultural worker; Take-home exposure
MeSH Terms: conditions — Dehydration; Heat Stress Disorders | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All participants (Other): All participants will receive the intervention
  Interventions: Other: Education and resources provided by community health workers

INTERVENTIONS:
Other: Education and resources provided by community health workers — The intervention will consist of implementing existing tools provided by EPA's Design for the Environment program, CalOSHA and NIOSH sector-specific guidance for agricultural workers, the Imperial County Department of Public Health and materials from California Department of Toxics Substances Control. The investigators will utilize and adjust existing educational tools such as the Heat Illness Prevention plan developed by CalOSHA. In addition to the educational materials, the investigators will give each farmworker cooling working gear to be worn during their work-shift with (specialized clothes that has been used in other occupational settings). The investigators will provide all participants with a low-cost fan filter, known as Corsi-Rosenthal box built jointly by the community health/research team to reduce chemicals at home, and a small A/C unit to reduce heat stress.

SUMMARY:
The investigators are studying the dangers that farmworkers face while working in the fields and at home. The investigators goals are:

1. Measure how much heat and chemicals farmworkers in Imperial County are exposed to.

   The investigators will ask the participants to wear a special belt under their clothes during work to measure heat. The investigators will also put two small temperature monitors in the participant's home for a day. The investigators will collect a urine sample to check hydration, and also measure the participants height, weight, blood pressure, and some blood markers for diseases using a simple finger-prick test.

   To measure chemicals, the investigators will give the participants a wristband to wear for a week and hang another in the participants home. The investigators will also collect dust from each participant's home with a vacuum. Then, the investigators will analyze everything at San Diego State University.

   After collecting samples, a trained community health worker will ask the participants a few questions about their work, lifestyle, health symptoms, and any hazards they face. The investigators will meet the participants twice at their homes to distribute the tools which will later be collected. Once the tools are collected, the investigators will have the chance to follow up with the participants if they have any questions.
2. Provide help to lower heat and chemical exposure with the help of community health workers.
3. Measure heat and chemicals again using the same methods to see if the project made a difference.
4. Talk to participants about what they liked and how the investigators can make future projects better.

ELIGIBILITY:
Inclusion Criteria:

* Currently living in Imperial County, California, USA
* Currently work in agriculture
* Plan on living in Imperial Valley for the next 6 months

Exclusion Criteria:

* Not currently living in Imperial County, California, USA
* Not currently working in agriculture
* Not planning to live in Imperial Valley for the next 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-06-07 (Actual); Primary Completion 2025-12-15 (Actual); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Individual heat stress | Assessment at baseline (pre-intervention) and again immediately (week) after the intervention
  Skin temperature in degrees Celsius derived from skin temperature monitor worn against the participant's skin.
Participant household temperature | Assessment at baseline (pre-intervention) and again immediately (week) after the intervention
  Household temperature in degrees Celsius, derived from weather monitor placed in the participant's home.
Participant hydration level | Assessment at baseline (pre-intervention) and again immediately (week) after the intervention
  Specific gravity of participant's urine
Concentration of chemicals measured in silicon wristband worn by study participant | Assessment at baseline (pre-intervention) and again immediately (week) after the intervention
  Participants will be asked to wear a silicon wristbands twice; once at baseline and again after the intervention. The research team will collect the wristbands and transport them to San Diego State University for analysis of different classes of chemicals, including pesticides, organophosphates, pyrethroids, and legacy pollutants. The chemicals adhered to the wristbands will be extracted in ethyl acetate and then passed through a solid-phase extraction. Extracts will be analyzed using a two-dimensional gas chromatography coupled to time-of-flight mass spectrometry at San Diego State University. The final concentration of each chemical will be expressed as nanograms per gram of wristband.
Concentration of chemicals measured in silicon wristbands hung in the participant's household. | Assessment at baseline (pre-intervention) and again immediately (week) after the intervention
  Silicon wristbands will be hung in participants' homes twice; once at baseline and again after the intervention. The research team will collect the wristbands and transport them to San Diego State University for analysis of different classes of chemicals, including pesticides, organophosphates, pyrethroids, and legacy pollutants. The chemicals adhered to the wristbands will be extracted in ethyl acetate and then passed through a solid-phase extraction. Extracts will be analyzed using a two-dimensional gas chromatography coupled to time-of-flight mass spectrometry at San Diego State University. The final concentration of each chemical will be expressed as nanograms per gram of wristband.
Concentration of chemicals measured in participant's household dust collected with a vacuum | Assessment at baseline (pre-intervention) and again immediately (week) after the intervention
  The research team will visit the participant's home twice to collect the dust samples of the living area using a vacuum; once at baseline and again after the intervention. After collection, the research team will transport the dust samples to San Diego State University to measure the concentrations of different classes of chemicals, including pesticides, organophosphates, pyrethroids, and legacy pollutants. The chemicals in the dust will be extracted in ethyl acetate and then passed through a solid-phase extraction. Extracts will be analyzed using a two-dimensional gas chromatography coupled to time-of-flight mass spectrometry at San Diego State University. The final concentration of each chemical will be expressed as nanograms per gram of dust.

CONTACTS AND LOCATIONS:
Locations (1):
- Lideres Campesinas Imperial, El Centro, California, United States

IPD SHARING:
Plan to Share IPD: No